CLINICAL TRIAL: NCT02608853
Title: Estimation of Malignancy Rates Within Humedica Patient Populations Sampled to be Representative of Liraglutide Initiators and LEADER™ Trial Participants
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN2211-4259; U1111-1173-7000 (Other: WHO)
Record Dates: First submitted 2015-10-01; First posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Liraglutide-like Cohort
  Interventions: Other: No treatment given
- LEADER™-like Cohort
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No treatment is actively administered. Patients are treated according to routine clinical practice at the discretion of their treating physicians.

SUMMARY:
This study is conducted in the United States of America. The aim of this study is to estimate incidence rates of all malignant neoplasms, specific subgroups of malignant neoplasms, and acute pancreatitis among cohorts of antidiabetic drug users standardized to be representative of LEADER™ trial participants or liraglutide initiators within the Humedica Electronic Health Record (EHR) database.

ELIGIBILITY:
Inclusion Criteria:

* All Cohort Members: Members of each of the cohorts must have at least 12 months of baseline coverage within Humedica prior to the patients' index date (cohort- specific index dates are defined below). Within Humedica, baseline coverage will be defined as the date from the earliest observed encounter up to and including the index date. Patients must have at least 1 diagnosis of T2DM (250.X0 or 250.X2) prior to and including the date of the qualifying prescription, no prior diagnosis (inclusive of the index date) of T1DM (250.X1 or 250.X3) and no diagnosis of gestational diabetes within the previous 12 months (inclusive of the index date). Patients will not be eligible for inclusion if they have prior prescriptions for GLP-1 analogues (including liraglutide and exenatide) during the interval that would be considered the baseline period
* Liraglutide-like Cohort: To be eligible for inclusion in the Liraglutide-like Cohort, patients must have at least one qualifying prescription for an OAD. Qualifying OADs will be specified that share similar labelled or unlabelled indications as liraglutide
* LEADER™-like Cohort: To be eligible for inclusion in the LEADERTM-like Cohort, patients must meet the following inclusion and exclusion criteria: Patients will be eligible for inclusion after meeting the overall inclusion and exclusion criteria in addition to the following: Ages 50 and over. HbA1c at least 7%

Exclusion Criteria:

* Patients will be excluded from the LEADER™-like Cohort if any of the following are observed prior to meeting the inclusion criteria defined above: Calcitonin >= 50ng/L. Baseline DPP-4 or pramlintide. Chronic heart failure diagnosis, NYHA Class IV. Acute coronary or cerebrovascular event within 14 days prior to initiation. Current continuous renal replacement therapy. End-stage liver disease. Solid organ transplant. Malignant neoplasm

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include a cohort of patients with type 2 diabetes mellitus (T2DM) who initiated liraglutide and two cohorts of patients with T2DM standardized to have similar baseline covariates, including use of antidiabetic medicines, relative to the liraglutide initiators (the Liraglutide-like Cohort) and to participants in the LEADER™ Trial (LEADER™-like Cohort).
Sampling Method: Non-Probability Sample
Enrollment: 9999 (Actual)
Dates: Start 2015-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Incidence of all malignant neoplasms | Follow-up is defined as the period following the date of the qualifying prescription or diagnosis (01 Jan 2008 at the earliest) and will vary depending on when this date occurs. The follow-up study period ends on 31 Dec 2013 (in total up to 6 years)

SECONDARY OUTCOMES:
Incidence of specific malignant neoplasms - Breast (women only) | Follow-up is defined as the period following the date of the qualifying prescription or diagnosis (01 Jan 2008 at the earliest) and will vary depending on when this date occurs. The follow-up study period ends on 31 Dec 2013 (in total up to 6 years)
Incidence of specific malignant neoplasms - Colorectal | Follow-up is defined as the period following the date of the qualifying prescription or diagnosis (01 Jan 2008 at the earliest) and will vary depending on when this date occurs. The follow-up study period ends on 31 Dec 2013 (in total up to 6 years)
Incidence of specific malignant neoplasms - Pancreatic | Follow-up is defined as the period following the date of the qualifying prescription or diagnosis (01 Jan 2008 at the earliest) and will vary depending on when this date occurs. The follow-up study period ends on 31 Dec 2013 (in total up to 6 years)
Incidence of specific malignant neoplasms - Thyroid | Follow-up is defined as the period following the date of the qualifying prescription or diagnosis (01 Jan 2008 at the earliest) and will vary depending on when this date occurs. The follow-up study period ends on 31 Dec 2013 (in total up to 6 years)
Incidence of specific malignant neoplasms - Medullary Thyroid | Follow-up is defined as the period following the date of the qualifying prescription or diagnosis (01 Jan 2008 at the earliest) and will vary depending on when this date occurs. The follow-up study period ends on 31 Dec 2013 (in total up to 6 years)
Incidence of acute pancreatitis | Follow-up is defined as the period following the date of the qualifying prescription or diagnosis (01 Jan 2008 at the earliest) and will vary depending on when this date occurs. The follow-up study period ends on 31 Dec 2013 (in total up to 6 years)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Clinical Trial Call Center, Princeton, New Jersey, United States

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com